CLINICAL TRIAL: NCT00335959
Title: Neoadjuvant Chemoradiation Therapy With Oxaliplatin and Capecitabine for Patients With Surgically Resectable Gastric Cancer: A Pilot Phase II Trial With Molecular Correlates
Brief Title: S0425 Oxaliplatin, Capecitabine, and RT in Treating Patients W/Stomach Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to slow accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000476577; U10CA032102 (NIH); S0425 (Other: SWOG)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-07

CONDITIONS: Gastric Cancer
Keywords: adenocarcinoma of the stomach; stage I gastric cancer; stage II gastric cancer; stage III gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin; Gastrectomy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy, Chemoradiation, Surgery (Experimental): Chemotherapy: Oxaliplatin, 130 mg/m2, 2 hour IV infusion on Days 1 and 22; Capecitabine 850 mg/m2/dose, PO q 12 hours on Days 1-14 and 22-35 Chemoradiation: Capecitabine 650 mg/m2/dose, PO q 12 hours on days 43-77; Radiation therapy 180 cGy/day, 5 days/week beginning on Day 43.
  Surgery: Distal subtotal gastrectomy, total gastrectomy, or proximal gastrectomy
  Interventions: Drug: capecitabine; Drug: oxaliplatin; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: capecitabine — 850 mg/m2/dose PO q 12 hours Days 1-14 and 22-35. 650 mg/m2/dose PO q 12 hours Days 43-77.
  Other Names: Xeloda (NSC-712807)
Drug: oxaliplatin — 130 mg/m2 by 2-hour infusion Days 1 and 22
  Other Names: Eloxatin (NSC-266046)
Procedure: conventional surgery — Distal subtotal gastrectomy, total gastrectomy, or proximal gastrectomy
  Other Names: gastrectomy
Radiation: radiation therapy — Beginning Day 43, patients will be treated 5 days/week at 180 cGy/day times 25 fractions to a total dose of 4,500 cGy.
  Other Names: RT

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving oxaliplatin and capecitabine together with radiation therapy works in treating patients with stomach cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pathologic complete response rate in patients with primary gastric adenocarcinoma treated with neoadjuvant chemoradiotherapy comprising oxaliplatin, capecitabine, and radiotherapy. (This will not be completed as this study was closed early due to poor accrual.)
* Assess the frequency and severity of toxicities associated with this regimen.
* Explore, preliminarily, the association between DNA repair genes (ERCC-1, XRCC1, GST-P1, XPD, XPA, ribonucleotide reductase), target enzymes (thymidylate synthase [TS], dihydropyrimidine dehydrogenase, thymidine phosphorylase [TP]), and angiogenic factors (vascular endothelial growth factor [VEGF], epidermal growth factor [EGF], PD-ECGF, basic fibroblast growth factor, TSP-1 and -2, transforming growth factor [TGF]-β, and IL-8) and response to neoadjuvant therapy in patients with adenocarcinoma of the stomach. (This will not be completed as this study was closed early due to poor accrual.)
* Explore, preliminarily, the association of haplotypes of candidate genes of TS, TP, ERCC-1, XPD, GST-P1, cyclooxygenase-2, EGF receptor, TGF-β, VEGF, and IL-8 with response and toxicity to neoadjuvant chemoradiation therapy in these patients. (This will not be completed as this study was closed early due to poor accrual.)
* Explore, preliminarily, the feasibility of performing comparative genomic hybridization for analysis of DNA copy number changes in predicting response to neoadjuvant chemoradiation therapy. (This will not be completed as this study was closed early due to poor accrual.)

OUTLINE: This is a multicenter, pilot study.

* Neoadjuvant chemotherapy: Patients receive oxaliplatin IV over 2 hours on days 1 and 22 and oral capecitabine twice daily on days 1-14 and 22-35 in the absence of disease progression or unacceptable toxicity.
* Neoadjuvant chemoradiotherapy: Patients receive oral capecitabine twice daily on days 43-77 and undergo radiotherapy once daily on days 43-47, 50-54, 57-61, 64-68, and 71-75 in the absence of disease progression or unacceptable toxicity.
* Surgery: Patients with stable or responding disease undergo surgery 4-6 weeks after completion of chemoradiotherapy.

Tumor tissue is obtained at surgery or endoscopic biopsy. Gene expression analysis and comparative genomic hybridization testing are conducted on the tissue. Blood is drawn prior to beginning study treatment and is analyzed for germline polymorphisms.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary adenocarcinoma of the stomach, meeting the following criteria:

  * Newly diagnosed disease amenable to curative resection
  * Stage IB-III (T2-4)
* Measurable or nonmeasurable disease
* Enlarged lymph nodes outside of radiation fields must have preoperative biopsies

  * No positive lymph nodes outside of radiation fields
* No distant metastasis
* No gastroesophageal junction tumors

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* WBC ≥ 3,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal
* Albumin ≥ 3 g/dL
* Bilirubin normal
* No evidence of ischemic heart disease by EKG
* No coronary artery disease requiring active medical treatment
* No symptoms of angina
* No history of myocardial infarction
* No deep vein thrombosis within the past 12 months
* No pre-existing peripheral neuropathy
* No active pneumonia or inflammatory lung infiltrate
* No prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for ≥ 5 years
* No clinically significant comorbid medical conditions that would prevent delivery of chemotherapy, radiotherapy, or the performance of surgery
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior and no concurrent sorivudine or brivudine
* No prior therapy for this malignancy, including chemotherapy, surgery, immunotherapy, or radiotherapy
* No prior coronary angioplasty or stenting
* No concurrent 2-dimensional or intensity-modulated radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P. Leichman, MD, Study Chair — Desert Regional Medical Center Comprehensive Cancer Center; Syed A. Ahmad, MD, Study Chair — Barrett Cancer Center
Locations (75):
- United States (75):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy, Chemoradiation, Surgery: Oxaliplatin 130 mg/m2 (2 hour IV infusion on Days 1 and 22), Capecitabine 850 mg/m2/dose (PO q 12 hours on Days 1-14 and 22-35), Capecitabine 650 mg/m2/dose (PO q 12 hours on days 43-77), Radiation therapy 180 cGy/day, 5 days/week beginning on Day 43. Patients with stable disease or better were to have distal subtotal gastrectomy, total gastrectomy, or proximal gastrectomy.
Period: Overall Study
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Started | 7
Eligible | 6
Eligible and Began Protocol Therapy | 6
Completed | 4
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 6
Age Continuous [Median (Full Range); unit: years] — All eligible patients were included in this measure.
  years | 72 [29.8 to 86.9]
Sex: Female, Male [Count of Participants; unit: Participants] — All eligible patients were included in this measure.
  Participants
    Female | 3
    Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All eligible patients were included in this measure.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 3
    Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — All eligible patients were included in this measure.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 3
    More than one race | 0
    Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5= Fatal.
Time Frame: Patients were assessed for adverse events after pre-operative chemotherapy, after pre-operative chemoradiation and within 14 days of surgery.
Population: Eligible patients who received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants with a given type of AE
Groups:
- Chemotherapy, Chemoradiation and Surgery: Patients were to receive Oxaliplatin 130 mg/m2 (2 hour IV infusion on Days 1 and 22), Capecitabine 850 mg/m2/dose (PO q 12 hours on Days 1-14 and 22-35), Capecitabine 650 mg/m2/dose (PO q 12 hours on days 43-77), Radiation therapy 180 cGy/day, 5 days/week beginning on Day 43. Patients with stable disease or better were to have distal subtotal gastrectomy, total gastrectomy, or proximal gastrectomy.
Arm/Group | Chemotherapy, Chemoradiation and Surgery
Number analyzed (Participants) | 6
Participants with a given type of AE
  Anorexia | 1
  Dehydration | 2
  Diarrhea | 2
  Fatigue (asthenia, lethargy, malaise) | 1
  Gastrointestinal-Other (Specify) | 1
  Hemoglobin | 1
  Leukocytes (total WBC) | 1
  Lymphopenia | 2
  Nausea | 1
  Necrosis, GI - Small bowel NOS | 1
  Neutrophils/granulocytes (ANC/AGC) | 1
  Phosphate, serum-low (hypophosphatemia) | 1
  Platelets | 1
  Potassium, serum-low (hypokalemia) | 1
  Sodium, serum-low (hyponatremia) | 1
  Vomiting | 1

2. Primary Outcome: Pathologic Complete Response
Description: Pathologic complete response rates (pCR) of primary gastric adenocarcinoma when treated with oxaliplatin and capecitabine followed by capecitabine and radiation pre-operatively. On review of the resected gastric specimen and accompanying lymph nodes, pCR is no cancer recognized by the pathologist. Margins are free of tumor.
Time Frame: 17-19 weeks
Population: Eligible patients who completed pre-operative therapy were assessed for response.
Measure: Number; unit: participants
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 5
participants
  Unconfirmed Complete Response | 1
  Unconfirmed Partial Response | 2
  Stable/No Response | 2
  Increasing Disease | 1
  Assessment Inadequate | 1

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events after pre-operative chemotherapy, after pre-operative chemoradiation and within 14 days of surgery.
Arm/Group | Chemotherapy, Chemoradiation and Surgery
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy, Chemoradiation and Surgery (N=6)
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy, Chemoradiation and Surgery (N=6)
Hemoglobin (Blood and lymphatic system disorders) | 4
Ventricular arrhythmia - PVCs (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Necrosis, GI - Small bowel NOS (Gastrointestinal disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - Esophagus (Gastrointestinal disorders) | 1
Pain - Intestine (Gastrointestinal disorders) | 1
Pain - Stomach (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Urinary tract (Infections and infestations) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
Creatinine (Investigations) | 2
Leukocytes (total WBC) (Investigations) | 4
Lymphopenia (Investigations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Platelets (Investigations) | 2
Weight loss (Investigations) | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 4
Mood alteration - anxiety (Psychiatric disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No